CLINICAL TRIAL: NCT03987737
Title: Rectal Gas Removal Through Small Catheter Placement Prior to MRI of the Prostate: Assessment of the Impact on Diffusion Weighted Images Artifacts and Diagnostic Accuracy
Brief Title: Rectal Gas Removal Through Small Catheter Placement Prior to MRI of the Prostate
Acronym: GAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: s.-nr
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Prostatic neoplasm; Prostate; bp MRI of the prostate; small rectal catheter placement
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, comparative study between two rectal emptying strategies. Patients will be randomized into one of two arms. In both arms the subjects will be asked to evacuate the rectum as much as possible prior to the MRI exam. In the study arm, a small catheter will be placed in the rectum by the MRI technician and the examination will be executed with the small catheter in situ. In the control arm, subjects will be scanned immediately after rectal evacuation on the toilet. If the DWI sequence is non-interpretable due to susceptibility artefacts, excessive air will be removed with small catheter placement eventually and the scan will be repeated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- small catheter (Experimental): In the study arm, a small catheter will be placed in the rectum by the MRI technician and the examination will be executed with the small catheter in situ.
  Interventions: Procedure: small urinary catheter placement in the rectum
- control group (No Intervention): In the control arm, subjects will be scanned immediately after rectal evacuation on the toilet without small catheter in situ.

INTERVENTIONS:
Procedure: small urinary catheter placement in the rectum — The MRI technician will place a small urinary catheter in the rectum prior to MRI of the prostate to evacuate excessive gasses. This catheter will stay in the rectum during the whole MRI examination.
  Arms: small catheter

SUMMARY:
The presence of rectal gas can cause distortion at air-tissue interfaces on diffusion-weighted images (DWI) of prostate MRI and reduce image quality due to these susceptibility artifacts. Small catheter placement in the rectum before MRI is one of the ways that is advocated in PI-RADS v2 guidelines to reduce rectal gas. The goal of this study is to prospectively evaluate the effect of small catheter placement on artifacts on diffusion weighted images and to see whether it improves diagnostic accuracy.

DETAILED DESCRIPTION:
The value of MRI in the detection of clinically significant prostate cancer has already been shown in many studies [1]. With MRI widely available and general accepted by urologists and radiologist for prostate imaging, a good execution and high quality of the images have become crucial. Recently Caglic et al published an article about optimizing prostate mpMRI [2]. One of the factors that influences image quality is rectal loading and bowel movement. The prostate is located anterior in the immediate vicinity of the rectum, so prostatic MRI is prone to artifacts caused by bowel movements and to susceptibility artifacts at the air-tissue interface [3]. Rectal movements are correlated to the degree of rectal distension and result in significant displacement of the prostate gland [4]. Rectal distension has a negative impact on the quality of both T2-weighted (T2W) and diffusion weighted images (DWI) [5], which are the two most important sequences in the detection of clinically significant prostate cancer. A study by Lim et al [6] showed a significant correlation between the amount of stool in the rectum and the severity of motion artifacts, however reducing the amount of stool with an enema did not improve the quality of T2W, DWI or dynamic contrast enhanced (DCE) images compared to the non-enema group. As the authors have declared, this could be due to the fact that only a minority of patients in the non-enema group had moderate or large amounts of stool (15.6%).

This study by Lim et al also showed that the amount of rectal gas did not correlate with the severity of distortion artifacts on diffusion images, which could mean that even a small amount of gas could already cause substantial (susceptibility) artifacts on DWI. A larger study by Griethuysen et al [7] showed that a micro-enema shortly before the examination reduces both the incidence and the severity of gas-induced artifacts.

So, moving gas appears to be the main concern and preparation is recommended. There is no evidence that one rectal emptying strategy is better than another [8]. In PI-RADS v2, different approaches are suggested, the aforementioned micro-enema, performing the MRI exam with patient in the prone position or to decompress the rectum using a small catheter [9].

This study aims to assess the efficacy of small catheter placement just before the MRI examination in reducing susceptibility on diffusion weighted images.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study by giving written informed consent.
* male subjects aged between 45 to 80 years.
* scheduled for a prostate MRI due to clinical suspicion of prostatic carcinoma (elevated prostate specific antigen (PSA) levels in blood and/or abnormal digital rectal examination (DRE)), staging, follow-up or active surveillance.
* good health condition based on medical history, physical examination and vital sign measurements.

Exclusion Criteria:

* has a contra-indication for MRI (claustrophobia, non-compatible metallic implants).
* has a prior history of hip prosthesis.
* has any condition, physical, mental, familial or sociological, that could impede compliance with the study protocol and further follow-up. This is not an absolute contra-indication, but should be discussed with patient prior to registration in the trial.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participants needs to have a prostate
Enrollment: 46 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
degree of distortion of the prostate on AP direction on DWI compared to T2W images in mm | 1 week
  The difference in diameter in anterio-posterior direction between axial DWI and the corresponding T2W images

SECONDARY OUTCOMES:
Number of clinically significant cancers detected more due to improved quality of images | within 1 year
  compared to control group, and with biopsy/pathological specimen as reference
Number of rescans due to insufficient image quality after small catheter placement | within 1 year
  compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Mai, MD, Principal Investigator — University Hospital Leuven, Department of Radiology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Futterer JJ, Briganti A, De Visschere P, Emberton M, Giannarini G, Kirkham A, Taneja SS, Thoeny H, Villeirs G, Villers A. Can Clinically Significant Prostate Cancer Be Detected with Multiparametric Magnetic Resonance Imaging? A Systematic Review of the Literature. Eur Urol. 2015 Dec;68(6):1045-53. doi: 10.1016/j.eururo.2015.01.013. Epub 2015 Feb 2. PMID 25656808
- [Result] Caglic I, Barrett T. Optimising prostate mpMRI: prepare for success. Clin Radiol. 2019 Nov;74(11):831-840. doi: 10.1016/j.crad.2018.12.003. Epub 2019 Jan 2. PMID 30611559
- [Result] Mazaheri Y, Vargas HA, Nyman G, Akin O, Hricak H. Image artifacts on prostate diffusion-weighted magnetic resonance imaging: trade-offs at 1.5 Tesla and 3.0 Tesla. Acad Radiol. 2013 Aug;20(8):1041-7. doi: 10.1016/j.acra.2013.04.005. PMID 23830610
- [Result] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Result] Caglic I, Hansen NL, Slough RA, Patterson AJ, Barrett T. Evaluating the effect of rectal distension on prostate multiparametric MRI image quality. Eur J Radiol. 2017 May;90:174-180. doi: 10.1016/j.ejrad.2017.02.029. Epub 2017 Feb 22. PMID 28583630
- [Result] Lim C, Quon J, McInnes M, Shabana WM, El-Khodary M, Schieda N. Does a cleansing enema improve image quality of 3T surface coil multiparametric prostate MRI? J Magn Reson Imaging. 2015 Sep;42(3):689-97. doi: 10.1002/jmri.24833. Epub 2014 Dec 30. PMID 25556957
- [Result] van Griethuysen JJM, Bus EM, Hauptmann M, Lahaye MJ, Maas M, Ter Beek LC, Beets GL, Bakers FCH, Beets-Tan RGH, Lambregts DMJ. Gas-induced susceptibility artefacts on diffusion-weighted MRI of the rectum at 1.5 T - Effect of applying a micro-enema to improve image quality. Eur J Radiol. 2018 Feb;99:131-137. doi: 10.1016/j.ejrad.2017.12.020. Epub 2017 Dec 28. PMID 29362144
- [Result] McNair HA, Wedlake L, Lips IM, Andreyev J, Van Vulpen M, Dearnaley D. A systematic review: effectiveness of rectal emptying preparation in prostate cancer patients. Pract Radiat Oncol. 2014 Nov-Dec;4(6):437-47. doi: 10.1016/j.prro.2014.06.005. Epub 2014 Aug 3. PMID 25407867